CLINICAL TRIAL: NCT04318275
Title: An Early Feasibility Study to Explore a Novel Objective Pain Measurement Using a Wearable Biosensor and a Novel Mobile Platform in Patients With Endometriosis (OPINE)
Brief Title: Objective Pain Measurement Using a Wearable Biosensor and a Mobile Platform in Patients With Endometriosis
Acronym: OPINE
Status: Completed | Type: Observational
Sponsor: Biofourmis Singapore Pte Ltd. (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: CT004-AMY004JG
Record Dates: First submitted 2019-12-22; First posted 2020-03-23 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
This study aims to explore a novel objective measurement for endometriosis-related pain. A variety of pain symptoms are associated with endometriosis, including dysmenorrhea, dyspareunia, dysuria, dyschezia and chronic pelvic pain. However, a clear characterization of pain typology and topology in populations with endometriosis, other gynecologic pathology, or a normal pelvis is lacking. Understanding the precise nature of the relationship between pain and endometriosis is important for the clinical management of affected women, given the body of evidence indicating that medical and surgical management for pain associated with endometriosis has been shown to be effective. Evaluating the relationship between pain and endometriosis, however, is challenging given that pain is difficult to measure and the mechanism by which endometriosis causes pain is not well understood. While previous studies have provided important data on the incidence of pelvic pain and endometriosis, little research has been done to assess both the typology and topology of pelvic pain, pain beyond the pelvis, endometriosis diagnosis, or severity of pain using operative findings and a standardized classification system.

DETAILED DESCRIPTION:
BACKGROUND ON ENDOMETRIOSIS

A variety of pain symptoms are associated with endometriosis, including dysmenorrhea, dyspareunia, dysuria, dyschezia and chronic pelvic pain. However, a clear characterization of pain typology and topology in populations with endometriosis, other gynecologic pathology, or a normal pelvis is lacking. Understanding the precise nature of the relationship between pain and endometriosis is important for the clinical management of affected women, given the body of evidence indicating that medical and surgical management for pain associated with endometriosis has been shown to be effective. Evaluating the relationship between pain and endometriosis, however, is challenging given that pain is difficult to measure and the mechanism by which endometriosis causes pain is not well understood. While previous studies have provided important data on the incidence of pelvic pain and endometriosis, little research has been done to assess both the typology and topology of pelvic pain, and pain beyond the pelvis, and endometriosis diagnosis and severity using operative findings and a standardized classification system.

Historically, pain has been measured using subjective scales to determine the presence of pain and its severity. Common scales include the numeric rating scale (NRS), visual analog scale (VAS), and visual response scale (VRS). While this is important information, self-reporting is a problematic metric for both diagnostic and research purposes as it depends on pain history, cognitive and behavioral factors, and can vary over time. Other measures used in clinical practice, such as the Biberoglu and Behrman (B&B) score, incorporate both patient and clinician assessments of pain. However, patients describe symptomatology and gynecologists evaluate tenderness and induration during physical examination with an exceedingly high risk of bias and inconsistent reproducibility. Over the past few years, significant advances have been made in the development of valid biomarkers or surrogate markers for the presence and severity of pain. Measurement of various physiology parameters like heart rate, heart rate variability and electrodermal activity have shown to be associated with the presence of pain and can aid clinical interpretation.

STUDY RATIONALE

Several ratings, such as the numeric rating scale (NRS) are mainly used in clinical trials to determine the presence and severity of pain associated with endometriosis. Patient Reported Outcomes (PRO) such as NRS can be problematic as they are subjective, containing recall bias, and can vary over time. Thus, a more accurate and objective measurement of pain is needed to evaluate the efficacy of treatment with pain associated with endometriosis.

ELIGIBILITY:
Inclusion criteria:

1. Able to give a written Informed Consent Form.
2. Patient who is willing to comply with study restrictions including E4® device management (wearing and charging the device) and Femme Rhythm Patient App Management (pairing E4® device and the patient Femme Rhythm App, and carrying the smartphone for answering questionnaires and data reporting)
3. Female patients aged ≥ 21 and < 50 years.
4. Patient who meets either A or B or both in the following criteria: A. Confirmed diagnosis of endometriosis (laparoscopy/laparotomy) performed WITHIN 10 YEARS prior to the study participation.

   B. Current clinical diagnosis (endometriotic cysts or deep infiltrating endometriosis detected by TVUS, TRUS or MRI) WITHIN 6 MONTHS prior to the study participation.
5. Patient who meets either A or B in the following criteria:

   A. Patient is NOT treated with hormonal agents for endometriosis WITHIN 4 WEEKS prior to study participation, and have regular menses (i.e. 21-38 days) within 38 days prior to the study participation.

   B. Patient started hormonal agents for endometriosis, including combined oral contraceptives MORE THAN 8 WEEKS prior to the study participation, or progestins, danazol, GnRH agonists, GnRH antagonists or Progesterone and Levonorgestrel Releasing IUDs MORE THAN 12 WEEKS prior to the study participation, AND stable use of the medication is expected during the study period
6. Patient has a moderate to severe endometriosis- associated pelvic pain using the Monthly Assessment of Endometriosis Pain within 28 days prior to study participation

Exclusion criteria:

1. Patient is pregnant, or breast feeding or is planning a pregnancy during participation of the study or is less than 6 months postpartum, post-abortion, or post-pregnancy before participation.
2. Patient has chronic pelvic pain that is not caused by endometriosis that requires chronic analgesic or other chronic therapy, or that would interfere with the assessment of endometriosis related pain (e.g., pelvic inflammatory disease).
3. Patient has more than five surgical histories in pelvic area.
4. Patient has a skin disease or condition that would interfere with the collection or interpretation of physiological data obtained through E4®
5. Patient required neuromodulator (a long-acting or immediate release narcotic, or gabapentin) during 3 months prior to the study participation.
6. Patient has a planned surgery during the study.
7. Patient had a surgery within 4 weeks prior to the study participation.
8. Patient has a planned trip overseas during the study participation.
9. Any other reason that, in the judgment of the investigator, would render the subject unsuitable for the study participation.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female on self-representation and confirmed diagnosis of endometriosis by TVUS or MRI.
Study Population: 124 study participants, aged between 21 to 50 years old, female, who is confirmed diagnosis of endometriosis.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
The concordance between Pain Index and NRS scores during the study period. (Categorised into none, mild, moderate and severe pain) | 12 weeks
  Pain Index will be generated via vital sign collected from subjects and processed by Biofourmis's propriety algorithm. Both pain index and NRS will be categorised into None (0), Mild (1-3), Moderate (4-6), and Severe (7-10) pain.
  Concordance will be measured using unweighted Kappa Statistic for multiple categories with 95% CI. Percentage agreement between the categories will be also calculated by taking the number of concordant pairs divided by the total number of pain episodes.

SECONDARY OUTCOMES:
The correlation between 11-point Pain Index (0-10) and 11-point NRS score (0-10). | 12 weeks
  The generated Pain Index will be classified into 11 points (0-10) in accordance with the raw NRS score.
  Correlation between the 11-point Pain Index and raw NRS score will be measured using Spearman correlation.

OTHER OUTCOMES:
Exploratory Endpoint 1: Correlation between Quality of Life (EQ-5D-5L and EHP-30), Productivity (HRPQ), PROMIS-Fatigue with Sleep Quality and Stress Values calculated using Biofourmis's propriety algorithm. | 12 weeks
  The Pearson correlation and its statistical significance between the various Quality of Life measures and the Sleep Quality and Stress Values (calculated using Biofourmis's propriety algorithm) will be presented in a matrix table.
Exploratory Endpoint 2: Trend of Quality of Life over the study period | 12 weeks
  The trend of Quality of life measures will be presented using line charts.
Exploratory Endpoint 3: Trend of Pain Index and NRS categories over the study period | 12 weeks
  The trend of Pain Index and NRS categories (None, Mild, Moderate, Severe) will be presented using bar graphs.
Exploratory Endpoint 4: Effect of concomitant medication usage on the NRS categories | 12 weeks
  Effects of concomitant medication usage will be measured as an increment or decrement in NRS pain categories (None, Mild, Moderate, Severe), based on the highest pain reported by patient before taking the medication and the pain report after medication usage.
Exploratory Endpoint 5: Effect of concomitant medication usage on the Pain Index categories | 12 weeks
  Effects of concomitant medication usage will be measured as an increment or decrement in Pain Index categories (None, Mild, Moderate, Severe), based on the highest pain reported by patient before taking the medication and the Pain Index generated based on the pain report after medication usage.
Exploratory Endpoint 6: Correlation between EQ-5D-5L and physiological parameters. | 12 weeks
  The correlation between EQ-5D-5L and physiological parameters will be presented as scatterplots with the Pearson correlation and statistical significance.
Exploratory Endpoint 7: Correlation between EHP-30 and physiological parameters. | 12 weeks
  The correlation between EHP-30 and physiological parameters will be presented as scatterplots with the Pearson correlation and statistical significance.
Exploratory Endpoint 8: Correlation between Productivity (HRPQ) and physiological parameters. | 12 weeks
  The correlation between Productivity (HRPQ) and physiological parameters will be presented as scatterplots with the Pearson correlation and statistical significance.
Exploratory Endpoint 9: Correlation between PROMIS-Fatigue and physiological parameters. | 12 weeks
  The correlation between PROMIS-Fatigue and physiological parameters will be presented as scatterplots with the Pearson correlation and statistical significance.
Exploratory Endpoint 10: Change in Pain Index, NRS categories over the menstrual cycle. | 12 weeks
  Changes in Pain Index, NRS categories (None, Mild, Moderate, Severe) over the menstrual cycle will be summarized by plotting bar graphs across menstrual cycle.
Exploratory Endpoint 11: Change in physiological parameters over the menstrual cycle. | 12 weeks
  Changes in physiological parameters over the menstrual cycle will be summarized using boxplots across menstrual cycle.
Exploratory Endpoint 12: Change in Pain Index, NRS categories by the type of lesions | 12 weeks
  Changes in Pain Index, NRS categories (None, Mild, Moderate, Severe) over the lesion types will be summarized using bar graphs across the menstrual cycle.
Exploratory Endpoint 13: Change in physiological parameters by the type of lesions | 12 weeks
  Changes in physiological parameters over the lesion types will be summarized using boxplots across the menstrual cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Maulik Majmudar, M.D., Study Chair — Biofourmis Inc.
Locations (7):
- United States (2):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Rochester, Minnesota
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fauconnier A, Chapron C. Endometriosis and pelvic pain: epidemiological evidence of the relationship and implications. Hum Reprod Update. 2005 Nov-Dec;11(6):595-606. doi: 10.1093/humupd/dmi029. Epub 2005 Sep 19. PMID 16172113
- [Background] Ballard KD, Seaman HE, de Vries CS, Wright JT. Can symptomatology help in the diagnosis of endometriosis? Findings from a national case-control study--Part 1. BJOG. 2008 Oct;115(11):1382-91. doi: 10.1111/j.1471-0528.2008.01878.x. Epub 2008 Aug 19. PMID 18715240
- [Background] Cox L, Ayers S, Nala K, Penny J. Chronic pelvic pain and quality of life after laparoscopy. Eur J Obstet Gynecol Reprod Biol. 2007 Jun;132(2):214-9. doi: 10.1016/j.ejogrb.2006.04.020. Epub 2006 May 30. PMID 16730874
- [Background] Kang SB, Chung HH, Lee HP, Lee JY, Chang YS. Impact of diagnostic laparoscopy on the management of chronic pelvic pain. Surg Endosc. 2007 Jun;21(6):916-9. doi: 10.1007/s00464-006-9047-1. Epub 2006 Nov 14. PMID 17103271
- [Background] Ballard K, Lane H, Hudelist G, Banerjee S, Wright J. Can specific pain symptoms help in the diagnosis of endometriosis? A cohort study of women with chronic pelvic pain. Fertil Steril. 2010 Jun;94(1):20-7. doi: 10.1016/j.fertnstert.2009.01.164. Epub 2009 Apr 1. PMID 19342028
- [Background] Hsu AL, Sinaii N, Segars J, Nieman LK, Stratton P. Relating pelvic pain location to surgical findings of endometriosis. Obstet Gynecol. 2011 Aug;118(2 Pt 1):223-230. doi: 10.1097/AOG.0b013e318223fed0. PMID 21775836
- [Background] Renner SP, Boosz AS, Burghaus S, Maihofner C, Beckmann MW, Fasching PA, Jud SM. Visual pain mapping in endometriosis. Arch Gynecol Obstet. 2012 Sep;286(3):687-93. doi: 10.1007/s00404-012-2369-4. Epub 2012 May 9. PMID 22569716
- [Background] Revised American Society for Reproductive Medicine classification of endometriosis: 1996. Fertil Steril. 1997 May;67(5):817-21. doi: 10.1016/s0015-0282(97)81391-x. No abstract available. PMID 9130884
- [Background] Bourdel N, Alves J, Pickering G, Ramilo I, Roman H, Canis M. Systematic review of endometriosis pain assessment: how to choose a scale? Hum Reprod Update. 2015 Jan-Feb;21(1):136-52. doi: 10.1093/humupd/dmu046. Epub 2014 Sep 1. PMID 25180023
- [Background] Yong PJ, Williams C, Bodmer-Roy S, Ezeigwe C, Zhu S, Arion K, Ambacher K, Yosef A, Wong F, Noga H, Britnell S, Yager H, Bedaiwy MA, Brotto LA, Albert AY, Lisonkova S, Allaire C. Prospective Cohort of Deep Dyspareunia in an Interdisciplinary Setting. J Sex Med. 2018 Dec;15(12):1765-1775. doi: 10.1016/j.jsxm.2018.10.005. Epub 2018 Nov 13. PMID 30446474
- [Background] Practice Committee of the American Society for Reproductive Medicine. Treatment of pelvic pain associated with endometriosis: a committee opinion. Fertil Steril. 2014 Apr;101(4):927-35. doi: 10.1016/j.fertnstert.2014.02.012. Epub 2014 Mar 13. PMID 24630080
- [Background] Rotondi MA, Donner A. A confidence interval approach to sample size estimation for interobserver agreement studies with multiple raters and outcomes. J Clin Epidemiol. 2012 Jul;65(7):778-84. doi: 10.1016/j.jclinepi.2011.10.019. Epub 2012 May 4. PMID 22560852
- [Background] Schliep KC, Mumford SL, Peterson CM, Chen Z, Johnstone EB, Sharp HT, Stanford JB, Hammoud AO, Sun L, Buck Louis GM. Pain typology and incident endometriosis. Hum Reprod. 2015 Oct;30(10):2427-38. doi: 10.1093/humrep/dev147. Epub 2015 Aug 11. PMID 26269529